CLINICAL TRIAL: NCT00791921
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group Trial to Assess the Efficacy, Pharmacokinetics, and Safety of CDP870 Without Coadministration of MTX in Japanese Active RA Patients in Whom MTX Cannot be Administrated.
Brief Title: Efficacy Confirmation Trial of CDP870 Without Coadministration of Methotrexate (MTX) in Japanese Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Collaborators: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDP870-275-08-003
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Results first posted 2012-08-06 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Certolizumab Pegol; Cimzia
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CDP870 200mg (Experimental): 400mg CDP870 given at Week0, 2, 4 and thereafter 200mg CDP870 given every 2weeks
  Interventions: Drug: CDP870
- Placebo (Placebo Comparator): Placebo of CDP870
  Interventions: Drug: Placebo of CDP870

INTERVENTIONS:
Drug: CDP870 — 400mg CDP870 given at Week0, 2, 4 and thereafter 200mg CDP870 given every 2weeks until Week22 subcutaneously(SC)
  Arms: CDP870 200mg
Drug: Placebo of CDP870 — Placebo given every 2 weeks until Week22 (SC)
  Arms: Placebo

SUMMARY:
The objectives of this study are to verify the superiority in efficacy (American College of Rheumatology 20%: ACR20) and investigate the pharmacokinetics and safety of CDP870 versus placebo without coadministration of MTX in active RA patients in whom MTX cannot be administrated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of adult-onset RA of at least 6 months but not longer than 15 years in duration as defined by the 1987 American College of Rheumatology classification criteria.
* Subjects must have active RA disease as defined by:

  * At least 6 tender joints and 6 swollen joints
  * ESR of 28 mm/hour or CRP of 2.0 mg/dL
* Subjects who have failed to respond or have been resistant to at least one DMARD (including MTX)
* Subjects in whom MTX cannot be administered for any of the reasons(incomplete response/safety concerns)

Exclusion Criteria:

* Patients who have a diagnosis of any other inflammatory arthritis
* Patients who have a secondary, non-inflammatory type of arthritis (eg, osteoarthritis, fibromyalgia)
* Patients who currently have, or who have a history of, a demyelinating or convulsive disease of the central nervous system (eg, multiple sclerosis, epilepsy)
* Patients who have NYHA (New York Heart Association) Class III or IV congestive heart failure
* Patients who currently have, or who have a history of, tuberculosis
* Patients who have a high risk of infection (with a current infectious disease, a chronic infectious disease, a history of serious infectious disease)
* Patients who currently have, or who have a history of, malignancy
* Female patients who are breastfeeding or pregnant, who are of childbearing potential
* Patients who previously received treatment with 2 or more anti-TNFα drugs or who previously failed to respond to treatment with 1 or more aint-TNFα drugs.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2008-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Chair — OPCJ
Locations (7):
- Japan (7):
  - Chube Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushuh Region
  - Shikoku Region

REFERENCES:
- [Derived] Yamamoto K, Takeuchi T, Yamanaka H, Ishiguro N, Tanaka Y, Eguchi K, Watanabe A, Origasa H, Iwai K, Sakamaki Y, van der Heijde D, Miyasaka N, Koike T. Efficacy and safety of certolizumab pegol without methotrexate co-administration in Japanese patients with active rheumatoid arthritis: the HIKARI randomized, placebo-controlled trial. Mod Rheumatol. 2014 Jul;24(4):552-60. doi: 10.3109/14397595.2013.843764. Epub 2013 Nov 1. PMID 24981319

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in Japan between 2008 and 2010.
Pre-assignment Details: Participant flow results are based on the safety set.
Period: Overall Study
Arm/Group | CDP870 200mg | Placebo
Started | 116 | 114
Completed | 82 | 18
Not Completed | 34 | 96
Not completed — Protocol planed | 24 | 88
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 8 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lack of study drug administration | 1 | 1
Not completed — Reason other than those above | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CDP870 200mg | Placebo | Total
Number analyzed (Participants) | 116 | 114 | 230
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 88 | 94 | 182
  >=65 years | 28 | 20 | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 56.0 (10.2) | 55.4 (9.8) | 55.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 88 | 171
  Male | 33 | 26 | 59
Region of Enrollment [Number; unit: participants]
  Japan | 116 | 114 | 230

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology 20% (ACR20) Response at Week 12
Description: ACR20 responders are subjects with at least 20% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1)Health Assessment Questionnaire-Disability Index (HAQ-DI), 2)C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGA-VAS)
Time Frame: Baseline, Week 12
Population: All 230 subjects (116 CDP 200 mg, 114 Placebo) included in the Full Analysis Set (FAS) are included in this analysis
Measure: Number; unit: percentage of participants
Arm/Group | CDP870 200mg | Placebo
Number analyzed (Participants) | 116 | 114
percentage of participants | 67.2 | 14.9
Statistical Analysis 1: Comparison: CDP870 200mg vs Placebo; For ACR20 responder rate at Week 12, comparison between the CDP870 200 mg group and the placebo group was performed; Test type: Superiority or Other; p < 0.05, Regression, Logistic

2. Secondary Outcome: American College of Rheumatology 20% (ACR20) Response at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: All 230 subjects (116 CDP 200 mg, 114 Placebo) included in the Full Analysis Set (FAS) are included in this analysis
Measure: Number; unit: percentage of participants
Arm/Group | CDP870 200mg | Placebo
Number analyzed (Participants) | 116 | 114
percentage of participants | 63.8 | 11.4
Statistical Analysis 1: Comparison: CDP870 200mg vs Placebo; Test type: Superiority or Other; p < 0.05, Regression, Logistic

ADVERSE EVENTS:
Time Frame: 24-week double blind phase, from Baseline to Week 24
Description: Of the 230 subjects in the Full Analysis Set (FAS), 230 are included in the adverse event reporting based upon the Safety Set (SS) population. The Safety Set includes all subjects randomized who received at least 1 dosing.
Arm/Group | CDP870 200mg | Placebo
Serious Adverse Events (participants affected / at risk) | 13/116 | 3/114
Other Adverse Events (participants affected / at risk) | 46/116 | 41/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDP870 200mg (N=116) | Placebo (N=114)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ileitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic dissection rupture (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDP870 200mg (N=116) | Placebo (N=114)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 4 (5) | 4 (4)
Nasopharyngitis (Infections and infestations) | 20 (23) | 16 (21)
Pharyngitis (Infections and infestations) | 6 (6) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 4 (4)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 14 (14)
Eczema (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 10 (11) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No